CLINICAL TRIAL: NCT01037361
Title: Cerebral Activity Related to Primary Motor Stereotypies in Children: An EEG Study
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100015; 10-N-0015
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-06-29

CONDITIONS: Movement Disorder
Keywords: Children and Adolescents; Motor Control; Movement-Related Potential; Stereotypic Movement Disorder; Electroencephalogram (EEG)
MeSH Terms: conditions — Movement Disorders; Stereotypic Movement Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Motor stereotypies are a movement disorder characterized by involuntary, repetitive, and rhythmic movements. These movements have a predictable pattern and seem purposeful, but they serve no obvious function, tend to be prolonged, and can be suppressed. Common examples of motor stereotypies include hand waving, head nodding, and body rocking.
* Researchers are interested in learning more about motor stereotypies. Many children with autism and other developmental disorders tend to exhibit these behaviors, but normal healthy children and even some adults have demonstrated motor stereotypies under certain conditions (including boredom and stress). More research is needed to determine the internal causes of and potential successful treatments for these behaviors.

Objectives:

- To use electroencephalography (EEG) to study cerebral activity related to stereotypies in children.

Eligibility:

- Children between 7 and 18 years of age who demonstrate stereotypy movements on a consistent basis (at least 10 times a day for at least 4 months).

Design:

* The study will require two visits to the National Institutes of Health Clinical Center.
* First visit: Outpatient screening visit to determine the child s eligibility for the study, including questionnaires for parents/guardians and a medical assessment of the stereotypies.
* Second visit: Participating children will spend 1 day in a room at the NIH Clinical Center Pediatric Day Hospital. During the visit, participants will wear a portable EEG unit to measure brain activity. For the first hour of the visit, researchers will perform movement tests to study the brain activity related to normal movements. For the rest of the day, participants may play games, watch television or movies, read, or nap, while continuing to wear the EEG to monitor brain activity related to the stereotypic movements.
* Participants will receive a small amount of compensation for their time and participation.

DETAILED DESCRIPTION:
Objective

Motor stereotypy is a common movement disorder observed in children and adolescents but whose pathophysiology is unknown. Therefore, our overall objective is to study cerebral activity related to stereotypies. First, we want to define whether motor stereotypies are preceded by a cortical potential, as it is observed before voluntary movements. We hypothesize that no pre-movement potentials will precede the stereotypies. However, if a pre-movement potential is observed, our secondary objective is to compare this potential to cortical potentials that precede voluntary movements. We also aim to study cortical potentials preceding voluntary movements in healthy children and to compare them with the potentials observed in children with stereotypies.

Study population

12 children presenting with primary motor stereotypies and 12 healthy children.

Design

Using 19 scalp electrodes, we will record the patients electroencephalographic (EEG) activity for up to 8 hours during one day. The electromyographic (EMG) activity of the muscles involved in the stereotypies will be recorded with surface EMG electrodes. Healthy children will undergo an EEG for 2 hours. During this EEG recording, they will be asked to perform arms movements.

Outcome measures

Primary outcomes: latency and amplitude of both evoked and induced activity (cortical potentials) related to motor stereotypies will be measured.

Secondary outcomes: latency and amplitude of evoked and induced activity related to voluntary movements will be measured.

ELIGIBILITY:
* Population

  12 children presenting with primary motor stereotypies will be recruited as well as 12 healthy children.

INCLUSION CRITERIA:

Patients:

Children will be eligible to participate if they meet the following criteria:

* Are 7 through 18 years old;
* Are identified as having complex-motor stereotypies with predominant movements consisting of repetitive arm flapping, hand waving, or finger wiggling movements (only children presenting with these movements will be included);
* Predominant stereotypic movements must have started before six years of age;
* Predominant stereotypic movements must have been present for at least four months and occur at least 10 times a day;
* Dr Harvey Singer must have witnessed movements either in person or via videotape.
* The use of medication that does not affect the central nervous system will be allowed during the study.
* Subjects with the diagnosis of ADHD, obsessive-compulsive disorder, conduct disorder, or learning disability can be included.

Healthy volunteers:

Children will be eligible to participate if they meet the following criteria:

* Are 7 through 18 years old;
* Are able to give informed assent.

EXCLUSION CRITERIA:

Patients:

Subjects will be excluded from this study if there is:

* Diagnosis of autism, autistic spectrum disorder, Asperger syndrome, Pervasive Developmental Disorder NOS, or mental retardation (IQ < 70);
* Concurrent significant medical, neurological, or psychiatric condition;

Use of tranquilizers, psychotropic drugs or medications which could modulate the cortical activity, or if subjects have taken these medications during the month prior to their screening visit. As a consequence, children under stimulant medications for ADHD will be excluded from the study.

Healthy volunteers:

* Abnormal neurological exam, current or past history of neurological disease or psychiatric disease. Patients with neurological diseases of the central nervous system that impair the motor system or cognitive function will be excluded;
* Use of tranquilizers, psychotropic drugs or medications which could modulate the cortical activity, or if subjects have taken these medications during the month prior to their screening visit.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2009-12-02; Study Completion 2012-06-29

PRIMARY OUTCOMES:
Latency and amplitude of evoked (ERPs) and induced (ERD) activity related to motor stereotypies.

SECONDARY OUTCOMES:
Measures of latency and amplitude of evoked and induced activity related to voluntary movements.

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Belluscio, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bodfish JW, Symons FJ, Parker DE, Lewis MH. Varieties of repetitive behavior in autism: comparisons to mental retardation. J Autism Dev Disord. 2000 Jun;30(3):237-43. doi: 10.1023/a:1005596502855. PMID 11055459
- [Background] Castellanos FX, Ritchie GF, Marsh WL, Rapoport JL. DSM-IV stereotypic movement disorder: persistence of stereotypies of infancy in intellectually normal adolescents and adults. J Clin Psychiatry. 1996 Mar;57(3):116-22. PMID 8617696
- [Background] Deecke L. Electrophysiological correlates of movement initiation. Rev Neurol (Paris). 1990;146(10):612-9. PMID 2263824